CLINICAL TRIAL: NCT03004469
Title: A Multicentre, Randomized, Double-blind, Parallel-group, Controlled Study, to Assess the Efficacy and Safety of P-3074 Cutaneous Spray, Solution, in the Treatment of Male Pattern Baldness
Brief Title: Study to Evaluate the Efficacy and Safety of P-3074 Topical Solution in the Treatment of Androgenetic Alopecia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Polichem S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PM1541
Record Dates: First submitted 2016-12-23; First posted 2016-12-28 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Alopecia, Androgenetic
MeSH Terms: conditions — Alopecia | interventions — Finasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- P-3074 + Finasteride Placebo (Experimental): Participants received topical application of P-3074 contained finasteride 0.25% in morning onto dry scalp only (up to 4 puffs) and followed by placebo of finasteride 1 milligram (mg) tablet orally once daily for 24 weeks.
  Interventions: Drug: P-3074; Drug: Finasteride Placebo
- P-3074 Vehicle + Finasteride Placebo (Placebo Comparator): Participants received topical application of P-3074 vehicle in morning onto dry scalp only (up to 4 puffs) and followed by placebo of finasteride 1 mg tablet orally once daily for 24 weeks.
  Interventions: Drug: P-3074 Vehicle; Drug: Finasteride Placebo
- Oral Finasteride + P-3074 Vehicle (Active Comparator): Participants received finasteride 1 mg tablet orally once daily followed by topical application of P-3074 vehicle in morning onto dry scalp only (up to 4 puffs) for the 24 weeks.
  Interventions: Drug: Finasteride; Drug: P-3074 Vehicle

INTERVENTIONS:
Drug: P-3074
  Other Names: finasteride topical solution
  Arms: P-3074 + Finasteride Placebo
Drug: Finasteride
  Other Names: Propecia
  Arms: Oral Finasteride + P-3074 Vehicle
Drug: P-3074 Vehicle
  Other Names: Vehicle of P-3074
  Arms: Oral Finasteride + P-3074 Vehicle; P-3074 Vehicle + Finasteride Placebo
Drug: Finasteride Placebo
  Other Names: Placebo of Finasteride
  Arms: P-3074 + Finasteride Placebo; P-3074 Vehicle + Finasteride Placebo

SUMMARY:
The purpose of this study is to confirm the clinical efficacy and the safety of P-3074 in participants with androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent before starting any study related procedures;
* Men 18 to 40 years of age;
* Men with mild to moderate vertex male pattern hair loss according to a modified Norwood/Hamilton classification scale (III vertex, IV or V);
* Participants willing to have a tattoo in the target area;
* Outpatients;
* Ability to comprehend the full nature and purpose of the study, including possible risks and side effects;
* Ability to co-operate with the Investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

* Clinically relevant abnormal skin scalp findings which could interfere with the aim of the study; in particular, abrasion, actinic keratosis, inflammatory disorders or any other abnormality;
* Participants who had had hair transplant surgery or hair weaving;
* Clinically relevant abnormal laboratory values indicative of physical illness;
* Ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study;
* History of local infections of skin and subcutaneous tissues of the head in the 3-months period before the trial inclusion;
* Relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases, that may interfere with the aim of the study;
* Suspicion of malignancy, including prostate cancer;
* History of infertility or difficulty fathering children;
* Participants who wish to conceive children during the study or whose sexual partner(s) is pregnant;
* Participants with active seborrheic dermatitis;
* History of varicocele;
* Concurrent use of systemic corticosteroids, topical corticosteroids in the balding area studied, anabolic steroids, or over-the-counter "hair restorers";
* Use of the following drugs with antiandrogenic properties within 6 months of study entry: flutamide, cyproterone acetate, estrogen, progesterone, cimetidine, spironolactone or ketoconazole;
* Participants who had been treated with any of the following drugs within the past year: minoxidil (topical or oral), zidovudine, cyclosporine, diazoxide, phenytoin, systemic interferon, psoralens, streptomycin, penicillamine, benoxaprofen, tamoxifen, phenothiazines or cytotoxic agents;
* Use of finasteride or dutasteride within previous 12 months;
* Light or laser treatment of scalp within previous 3 months;
* Participation in the evaluation of any drug for 3 months before this study, calculated from the first day of the month following the last visit of the previous study;
* History of drug, alcohol [>2 drinks/day defined according to USDA Dietary Guidelines 2010], caffeine (>5 cups coffee/tea/day) or tobacco abuse (10 cigarettes/day).

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 458 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Massana, MD, Study Director — Almirall, S.A.
Locations (46):
- Belgium (4):
  - Site #102, Brussels
  - Site #103, Brussels
  - Site #104, Brussels
  - Site #101, Ghent
- Germany (19):
  - Site #211, Augsburg
  - Site #202, Berlin
  - Site #212, Berlin
  - Site #216, Bochum
  - Site #210, Dresden
  - Site #217, Dresden
  - Site #221, Dresden
  - Site #203, Düsseldorf
  - Site #204, Freiburg im Breisgau
  - Site #206, Hamburg
  - Site #214, Hamburg
  - Site #218, Hamburg
  - Site #213, Hanover
  - Site #215, Karlsruhe
  - Site #220, Lübeck
  - Site #208, Münster
  - Site #219, Potsdam
  - Site #209, Schwerin
  - Site #201, Wuppertal
- Hungary (6):
  - Site #303, Budapest
  - Site #309, Budapest
  - Site #302, Debrecen
  - Site #308, Sátoraljaújhely
  - Site #301, Szolnok
  - Site #307, Szombathely
- Russia (9):
  - Site #401, Chelyabinsk
  - Site #402, Moscow
  - Site #407, Moscow
  - Site #411, Moscow
  - Site #409, Rostov
  - Site #403, Ryazan
  - Site #406, Saint Petersburg
  - Site #408, Saint Petersburg
  - Site #410, Yaroslavl
- Spain (8):
  - Site #503, Alicante
  - Site #505, Barakaldo
  - Site #502, Barcelona
  - Site #507, Córdoba
  - Site #501, Madrid
  - Site #504, Madrid
  - Site #508, Madrid
  - Site #506, Pamplona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in 5 countries, in 52 sites and initiated on 02 Aug 2016 (First participant first visit) and the study got completed on 05 Mar 2018 (Last participant last visit).
Pre-assignment Details: A total of 632 participants were screened, with 458 participants being randomized.
Groups:
- P-3074 + Finasteride Placebo: Participants received topical application of P-3074 contained finasteride 0.25% in morning onto dry scalp only (up to 4 puffs) and followed by placebo of finasteride 1-milligram (mg) tablet orally once daily for 24 weeks.
- Oral Finasteride + P-3074 Vehicle: Participants received finasteride 1 mg tablet orally once daily followed by topical application of P-3074 vehicle in morning onto dry scalp only (up to 4 puffs) for 24 weeks.
Period: Overall Study
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Started | 189 | 184 | 85
Completed | 128 | 135 | 60
Not Completed | 61 | 49 | 25
Not completed — Adverse Event | 6 | 4 | 6
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 23 | 14 | 6
Not completed — Non-Compliance with Study Drug | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Withdrawal by Subject | 29 | 27 | 10
Not completed — Other unspecified reason | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Population: The data presented here for the for all randomized participants in the study.
Groups:
- P-3074 + Finasteride Placebo: Participants received topical application of P-3074 contained finasteride 0.25% in morning onto dry scalp only (up to 4 puffs) and followed by placebo of finasteride 1mg tablet orally once daily for 24 weeks
- Total: Total of all reporting groups
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle | Total
Number analyzed (Participants) | 189 | 184 | 85 | 458
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.7 (5.4) | 32.0 (4.8) | 31.9 (5.6) | 31.9 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 189 | 184 | 85 | 458
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 0 | 3
  Black/African American | 0 | 0 | 1 | 1
  Caucasian/White | 187 | 181 | 83 | 451
  Other | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in Hair Growth Assessed by Target Area Hair Count (TAHC) in the Vertex at Week 24
Description: The change from baseline in the TAHC within a 1 cm^2 (square centimeter) of baldness area at Week 24, were assessed by macro photographic techniques analysis. The Investigator selected a target area in the anterior leading edge of the vertex thinning area. A small dot tattoo was placed in the center of the circle of the clipped hairs. Using the tattoo as a reference point, the circular area was photographed and a 1 cm^2 circular area within the target area was analysed. Change is the adjusted mean of Week 24 minus baseline.The analysis uses a covariance pattern model adjusted for treatment group, center, visit and treatment-by-visit interaction as fixed effects and baseline hair count as a covariate with an unstructured covariance structure.
Time Frame: Baseline and Week 24
Population: Intent-to-Treat (ITT) Population included all participants who had measurements both at baseline and on treatment: i.e. participants who had measurements in regards to hair count both at baseline and on treatment.
Measure: Mean (Standard Deviation); unit: Hairs
Groups:
- P-3074 + Finasteride Placebo: Participants received topical application of P-3074 contained finasteride 0.25% in morning onto dry scalp only (up to 4 puffs) and followed by placebo of finasteride 1 mg tablet orally once daily for 24 weeks.
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 105 | 97 | 48
Hairs | 20.2 (2.88) | 6.7 (3.01) | 21.1 (3.90)
Statistical Analysis 1: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Test type: Other; p < .001, Mixed linear model; LS Mean Difference = 13.6, 95% CI 2-sided [5.8 to 21.3], Standard Error of Mean 3.94

2. Secondary Outcome: Adjusted Mean Change From Baseline in Hair Growth Assessed by TAHC in the Vertex at Week 12
Description: The change from baseline in the TAHC within a 1 cm^2 of baldness area at Week 12, were assessed by macro photographic techniques analysis. The Investigator selected a target area in the anterior leading edge of the vertex thinning area. A small dot tattoo was placed in the center of the circle of the clipped hairs. Using the tattoo as a reference point, the circular area was photographed and a 1 cm^2 circular area within the target area was analysed. Change is the adjusted mean of Week 24 minus baseline.The analysis uses a covariance pattern model adjusted for treatment group, center, visit and treatment-by-visit interaction as fixed effects and baseline hair count as a covariate with an unstructured covariance structure.
Time Frame: Baseline and Week 12
Population: ITT Population included all participants who had measurements both at baseline and on treatment: i.e. participants who had measurements in regards to hair count both at baseline and on treatment.
Measure: Mean (Standard Deviation); unit: Hairs
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 105 | 97 | 48
Hairs | 20.4 (2.41) | 7.6 (2.46) | 22.5 (3.31)
Statistical Analysis 1: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Test type: Other; p < .001, Mixed linear model; LS Mean Difference = 12.8, 95% CI 2-sided [6.5 to 19.1], Standard Error of Mean 3.19

3. Secondary Outcome: Adjusted Mean Change From Baseline in Target Area Hair Width (TAHW) in the Vertex at Weeks 12 and 24
Description: The change from baseline in the TAHW within a 1 cm^2 of baldness area at Weeks 12 and 24, were assessed by macro photographic techniques analysis. The Investigator selected a target area in the anterior leading edge of the vertex thinning area. A small dot tattoo was placed in the center of the circle of the clipped hairs. Using the tattoo as a reference point, the circular area was photographed and a 1 cm^2 circular area within the target area was analysed. Change is the adjusted mean of Weeks 12 and 24 minus baseline, respectively.The analysis uses a covariance pattern model adjusted for treatment group, center, visit and treatment-by-visit interaction as fixed effects and baseline hair count as a covariate with an unstructured covariance structure.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Micrometer
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 105 | 97 | 48
Micrometer
  Week 12 | -1.1231 (0.30653) | -0.7207 (0.31033) | -0.6938 (0.41951)
  Week 24 | -0.8052 (0.35151) | -1.5289 (0.36691) | 0.7163 (0.46679)
Statistical Analysis 1: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Week 12; Test type: Other; p = 0.322, Mixed linear model; LS Mean Difference = -0.4024, 95% CI 2-sided [-1.2020 to 0.3971], Standard Error of Mean 0.40570
Statistical Analysis 2: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Week 24; Test type: Other; p = 0.131, Mixed linear model; LS Mean Difference = 0.7237, 95% CI 2-sided [-0.2184 to 1.6657], Standard Error of Mean 0.47799

4. Secondary Outcome: Adjusted Mean Overall Male Hair Growth Questionnaire (MHGQ) Score as Assessed by the Participant at Weeks 12 and 24
Description: Participants assessed their scalp hair using a validated, self-administered MHGQ, which was given in their language. The self-administered MHGQ overall score assessed using the following 5-point scale: 1 = very satisfied, 2 = satisfied, 3 = neutral (neither satisfied nor dissatisfied), 4 = dissatisfied, 5 = very dissatisfied. A higher score indicated a worse outcome. The questionnaire was administered to eligible participants to subjectively measure their perception of hair growth. A higher score indicated a worse outcome.
Time Frame: Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 105 | 97 | 48
score on a scale
  Week 12 | 2.9 (0.08) | 3.0 (0.09) | 2.8 (0.12)
  Week 24 | 2.8 (0.09) | 3.0 (0.10) | 2.9 (0.13)
Statistical Analysis 1: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Week 12; Test type: Other; p = 0.569, Mixed linear model; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.2], Standard Error of Mean 0.11
Statistical Analysis 2: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Week 24; Test type: Other; p = 0.129, Mixed linear model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.1], Standard Error of Mean 0.12

5. Secondary Outcome: Adjusted Mean Change From Baseline in Participants Hair Growth/Loss Assessed for the Vertex by Investigator at Weeks 12 and 24
Description: The local Investigator assessed change in hair growth from Baseline to Week 12 and from Baseline to Week 24, using a 7-point scale. The evaluation was done by the Investigator or designee, by comparing the global vertex view photograph obtained at baseline visit with the participants actual scalp at 12 and 24 weeks. For the purpose of assessment of changes in hair growth by Investigators screening visits (where global photos were taken) were used as Baseline. The change from Baseline in hair growth was assessed using the following 7-point scale: -3 = greatly decreased, -2 = moderately decreased, -1 = slightly decreased, 0 = no change, +1 = slightly increased, +2 = moderately increased, +3 = greatly increased. The analysis uses a covariance pattern model adjusted for treatment group, center, visit and treatment-by-visit interaction as fixed effects with an unstructured covariance structure.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 105 | 97 | 48
score on a scale
  Week 12 | 0.5 (0.10) | 0.4 (0.11) | 0.5 (0.15)
  Week 24 | 0.8 (0.09) | 0.3 (0.09) | 0.7 (12)
Statistical Analysis 1: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Week 12; Test type: Other; p = 0.708, Mixed linear model; LS Mean Difference = 0.1, 95% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Week 24; Test type: Other; p < .001, Mixed linear model; LS Mean Difference = 0.4, 95% CI 2-sided [0.2 to 0.7], Standard Error of Mean 0.12

6. Secondary Outcome: Adjusted Mean Change From Baseline in Participants Hair Growth/Loss at Weeks 12 and 24, Assessed for the Vertex by Blind Assessor
Description: An independent blinded assessor was responsible for evaluating, under blinded conditions, the screening global photographs of the target area for all participants. They evaluated the eligibility of each participants according to the clinical inclusion criteria. The independent blinded assessor assessed the change of the hair growth from Baseline to Week 12 and from Baseline to Week 24, using a 7-point scale: -3 = greatly decreased, -2 = moderately decreased, -1 = slightly decreased, 0 = no change, +1 = slightly increased, +2 = moderately increased, +3 = greatly increased. This assessment was performed by comparing the global photographs obtained at screening visit with those subsequently obtained at Weeks 12 and 24. The analysis uses a covariance pattern model adjusted for treatment group, center, visit and treatment-by-visit interaction as fixed effects with an unstructured covariance structure.
Time Frame: Baseline, Week 12 and Week 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 105 | 97 | 48
score on a scale
  Week 12 | 0.0 (0.08) | 0.2 (0.08) | 0.2 (0.11)
  Week 24 | 0.2 (0.09) | 0.1 (0.09) | 0.3 (0.12)
Statistical Analysis 1: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Week 12; Test type: Other; p = 0.179, Mixed linear model; LS Mean Difference = -0.1, 95% CI 2-sided [-0.3 to 0.1], Standard Error of Mean 0.10
Statistical Analysis 2: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Week 24; Test type: Other; p = 0.262, Mixed linear model; LS Mean Difference = 0.1, 95% CI 2-sided [-0.1 to 0.4], Standard Error of Mean 0.12

7. Secondary Outcome: Adjusted Mean International Index of Erectile Function (IIEF-2) Scores at Weeks 4, 8, 12 and 24
Description: The 15-question IIEF-2 Questionnaire (Sexual Function Questionnaire) was used to evaluate any changes in sexual function and activity, at Weeks 4, 8, 12 and 24. A score of 0-5 is awarded to each of the 15 questions that examine the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. Erectile function domain has 6 questions with the score for domain range from 0-30. Orgasmic function domain has 2 questions with the score for domain range from 0-10. , Sexual desire function domain has 2 questions with the score for domain range from 0-10. Intercourse satisfaction function domain has 3 questions with the score for domain range from 0-15. Overall Satisfaction domain has 2 questions with the score for domain range from 0-10. A higher score indicated a worse outcome in that domain.
Time Frame: Weeks 4, 8, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 105 | 97 | 48
score on a scale
  Erectile Function Score, Week 4 | 24.5 (0.76) | 26.2 (0.79) | 23.5 (1.08)
  Erectile Function Score, Week 8 | 24.3 (0.80) | 24.9 (0.83) | 24.4 (1.15)
  Erectile Function Score, Week 12 | 25.3 (0.73) | 25.5 (0.77) | 23.6 (1.04)
  Erectile Function Score, Week 24 | 25.3 (0.74) | 26.1 (0.79) | 24.9 (1.05)
  Orgasmic Function Score, Week 4 | 9.3 (0.21) | 9.0 (0.22) | 8.9 (0.30)
  Orgasmic Function Score, Week 8 | 8.7 (0.26) | 8.7 (0.27) | 9.1 (0.38)
  Orgasmic Function Score, Week 12 | 9.4 (0.21) | 8.9 (0.22) | 9.0 (0.30)
  Orgasmic Function Score, Week 24 | 8.9 (0.25) | 9.1 (0.26) | 9.0 (0.35)
  Sexual Desire Score, Week 4 | 7.3 (0.17) | 7.5 (0.17) | 7.1 (0.24)
  Sexual Desire Score, Week 8 | 7.4 (0.16) | 7.4 (0.17) | 7.6 (0.23)
  Sexual Desire Score, Week 12 | 7.7 (0.15) | 8.0 (0.16) | 7.8 (0.21)
  Sexual Desire Score, Week 24 | 7.7 (0.17) | 7.7 (0.18) | 7.8 (0.24)
  Intercourse Satisfaction Score, Week 4 | 9.4 (0.49) | 10.7 (0.51) | 8.5 (0.69)
  Intercourse Satisfaction Score, Week 8 | 9.6 (0.49) | 9.9 (0.51) | 9.0 (0.70)
  Intercourse Satisfaction Score, Week 12 | 9.9 (0.49) | 10.2 (0.51) | 8.3 (0.69)
  Intercourse Satisfaction Score, Week 24 | 9.8 (0.47) | 10.8 (0.50) | 8.9 (0.67)
  Overall Satisfaction Score, Week 4 | 7.9 (0.22) | 8.0 (0.22) | 7.9 (0.31)
  Overall Satisfaction Score, Week 8 | 7.9 (0.21) | 7.8 (0.22) | 7.8 (0.31)
  Overall Satisfaction Score, Week 12 | 8.1 (0.22) | 8.1 (0.23) | 7.6 (0.31)
  Overall Satisfaction Score, Week 24 | 8.0 (0.22) | 8.1 (0.23) | 8.2 (0.31)
Statistical Analysis 1: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Erectile Function Score, Week 4; Test type: Other; p = 0.103, Mixed linear model; LS Mean Difference = -1.7, 95% CI 2-sided [-3.7 to 0.3], Standard Error of Mean 1.03
Statistical Analysis 2: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Erectile Function Score, Week 8; Test type: Other; p = 0.545, Mixed linear model; LS Mean Difference = -0.7, 95% CI 2-sided [-2.8 to 1.5], Standard Error of Mean 1.10
Statistical Analysis 3: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Erectile Function Score, Week 12; Test type: Other; p = 0.842, Mixed linear model; LS Mean Difference = -0.2, 95% CI 2-sided [-2.2 to 1.8], Standard Error of Mean 1.0
Statistical Analysis 4: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Erectile Function Score, Week 24; Test type: Other; p = 0.449, Mixed linear model; LS Mean Difference = -0.8, 95% CI 2-sided [-2.8 to 1.2], Standard Error of Mean 1.02
Statistical Analysis 5: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Orgasmic Function Score, Week 4; Test type: Other; p = 0.272, Mixed linear model; LS Mean Difference = 0.3, 95% CI 2-sided [-0.2 to 0.9], Standard Error of Mean 0.28
Statistical Analysis 6: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Orgasmic Function Score, Week 8; Test type: Other; p = 0.918, Mixed linear model; LS Mean Difference = 0.0, 95% CI 2-sided [-0.7 to 0.8], Standard Error of Mean 0.36
Statistical Analysis 7: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Orgasmic Function Score, Week 12; Test type: Other; p = 0.078, Mixed linear model; LS Mean Difference = 0.5, 95% CI 2-sided [-0.1 to 1.1], Standard Error of Mean 0.078
Statistical Analysis 8: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Orgasmic Function Score, Week 24; Test type: Other; p = 0.593, Mixed linear model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.34
Statistical Analysis 9: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Sexual Desire Score, Week 4; Test type: Other; p = 0.295, Mixed linear model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.7 to 0.2], Standard Error of Mean 0.23
Statistical Analysis 10: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Sexual Desire Score, Week 8; Test type: Other; p = 0.926, Mixed linear model; LS Mean Difference = -0.0, 95% CI 2-sided [-0.5 to 0.4], Standard Error of Mean 0.22
Statistical Analysis 11: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Sexual Desire Score, Week 12; Test type: Other; p = 0.183, Mixed linear model; LS Mean Difference = -0.3, 95% CI 2-sided [-0.7 to 0.1], Standard Error of Mean 0.20
Statistical Analysis 12: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Sexual Desire Score, Week 24; Test type: Other; p = 0.981, Mixed linear model; LS Mean Difference = 0.0, 95% CI 2-sided [-0.4 to 0.5], Standard Error of Mean 0.23
Statistical Analysis 13: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Intercourse Satisfaction Score, Week 4; Test type: Other; p = 0.041, Mixed linear model; LS Mean Difference = -1.4, 95% CI 2-sided [-2.7 to -0.1], Standard Error of Mean 0.66
Statistical Analysis 14: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Intercourse Satisfaction Score, Week 8; Test type: Other; p = 0.562, Mixed linear model; LS Mean Difference = -0.4, 95% CI 2-sided [-1.7 to 0.9], Standard Error of Mean 0.67
Statistical Analysis 15: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Intercourse Satisfaction Score, Week 12; Test type: Other; p = 0.642, Mixed linear model; LS Mean Difference = -0.3, 95% CI 2-sided [-1.6 to 1.0], Standard Error of Mean 0.66
Statistical Analysis 16: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Intercourse Satisfaction Score, Week 24; Test type: Other; p = 0.156, Mixed linear model; LS Mean Difference = -0.9, 95% CI 2-sided [-2.2 to 0.4], Standard Error of Mean 0.65
Statistical Analysis 17: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Overall Satisfaction Score, Week 4; Test type: Other; p = 0.824, Mixed linear model; LS Mean Difference = -0.1, 95% CI 2-sided [-0.6 to 0.5], Standard Error of Mean 0.29
Statistical Analysis 18: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Overall Satisfaction Score, Week 8; Test type: Other; p = 0.713, Mixed linear model; LS Mean Difference = 0.1, 95% CI 2-sided [-0.5 to 0.7], Standard Error of Mean 0.29
Statistical Analysis 19: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Overall Satisfaction Score, Week 12; Test type: Other; p = 0.993, Mixed linear model; LS Mean Difference = 0.0, 95% CI 2-sided [-0.6 to 0.6], Standard Error of Mean 0.30
Statistical Analysis 20: Comparison: P-3074 + Finasteride Placebo vs P-3074 Vehicle + Finasteride Placebo; Statistical Analysis details presented here is for Overall Satisfaction Score, Week 24; Test type: Other; p = 0.550, Mixed linear model; LS Mean Difference = -0.2, 95% CI 2-sided [-0.8 to 0.4], Standard Error of Mean 0.30

8. Secondary Outcome: Local Tolerability as Assessed by Incidence Rate of Skin Irritation Event Via Severity Score for Skin Irritation Scale
Description: Local tolerability at the application site was assessed to rate the severity of any skin irritation. The Investigator used the Severity score for skin Irritation scale to assess local tolerability. The dermal response and other effects indicative irritation responses were recorded at time of examination. Anything other than "No evidence of irritation" under Dermal Response was considered as a Dermal Response Skin Irritation event. Anything other than "No other effects" under Other Effects was considered as an Other Effects of Skin Irritation event. The event incidence rate is calculated as the number of events interest divided by total personal time in years.
Time Frame: Baseline to Week 24
Population: Safety Population includes all randomized participants who received at least one application of the IMP.
Measure: Number; unit: Events per personal years
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 181 | 181 | 84
Events per personal years
  Dermal Response | 0.340 | 0.245 | 0.661
  Other Effects | 0.368 | 0.463 | 0.755

9. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An Adverse event is defined as any untoward medical occurrence in a participants or clinical investigation patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with treatment. A serious AE was an AE that results in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect and medically significant event. The Treatment Emergent Adverse Events (TEAEs) is defined as all AEs occurring on or after the first dose of the IMP.
Time Frame: From the start of IMP up to 28 weeks
Population: Safety Population includes all randomized participants who received at least one application of the IMP.
Measure: Number; unit: participants
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
Number analyzed (Participants) | 181 | 181 | 84
participants
  TEAEs | 75 | 76 | 41
  Serious TEAEs | 4 | 5 | 1

ADVERSE EVENTS:
Time Frame: From the start of the IMP up to 28 weeks
Description: The data presented here for the safety population which includes all randomized participants who receive at least one application of the IMP.
Arm/Group | P-3074 + Finasteride Placebo | P-3074 Vehicle + Finasteride Placebo | Oral Finasteride + P-3074 Vehicle
All-Cause Mortality (participants affected / at risk) | 0/181 | 0/181 | 0/84
Serious Adverse Events (participants affected / at risk) | 4/181 | 5/181 | 1/84
Other Adverse Events (participants affected / at risk) | 74/181 | 73/181 | 40/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P-3074 + Finasteride Placebo (N=181) | P-3074 Vehicle + Finasteride Placebo (N=181) | Oral Finasteride + P-3074 Vehicle (N=84)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Exposure via father (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Skull fractured base (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P-3074 + Finasteride Placebo (N=181) | P-3074 Vehicle + Finasteride Placebo (N=181) | Oral Finasteride + P-3074 Vehicle (N=84)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anal pruritus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Inguinal hernia perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Application site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 1 (2) | 1 (1)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatocellular injury (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Dust allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastritis helminthic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (4) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Infected bite (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 2 (2) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 28 (32) | 24 (29) | 15 (22)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pertussis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulpitis dental (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Testicular abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Crystal urine present (Investigations) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Liver function test increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Stress echocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cervicogenic headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (4) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 17 (25) | 20 (29) | 8 (9)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (2)
Burnout syndrome (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Initial insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Libido decreased (Psychiatric disorders) | 1 (1) | 3 (3) | 1 (1)
Loss of libido (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 2 (2)
Sexual dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal pruritus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (7) | 3 (3)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (3) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sebaceous gland disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
High risk sexual behaviour (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Stress at work (Social circumstances) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (4):
  • Study Protocol: Protocol Version 4 dated 8 Mar 2017 (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03004469/Prot_000.pdf
  • Study Protocol: Non-substantial amendment 1 dated 8 Mar 17 (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03004469/Prot_001.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan dated 22 Jan 2018 (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03004469/SAP_002.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan Amendment 1 dated 23 Mar 2018 (2018-03-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03004469/SAP_003.pdf